CLINICAL TRIAL: NCT04765111
Title: A Phase II Study of Acalabrutinib Plus Rituximab in Previously Untreated Elderly Patients With Mantle Cell Lymphoma
Brief Title: Acalabrutinib and Rituximab for the Treatment of Previously Untreated Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0858; NCI-2021-00538 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0858 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, rituximab) (Experimental): Patients receive acalabrutinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV over 3-4 hours on days 1, 8, 15, and 22 of cycle 1, and day 1 of cycles 2-12, 14, 18, 20, 22, and 24. Cycles repeats every 28 days for up to 24 months or until complete remission is achieved in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Biological: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies the side effects of acalabrutinib and rituximab and its effect in treating patients with previously untreated mantle cell lymphoma. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that binds to a protein called CD20, which is found on B-cells, and may kill cancer cells. Giving acalabrutinib and rituximab may help to control mantle cell lymphoma in elderly patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy measured by complete remission (CR) rate of the acalabrutinib in combination with rituximab in newly diagnosed elderly mantle cell lymphoma (MCL) patients.

II. To determine the safety profile of acalabrutinib with rituximab combination in elderly patients with MCL.

SECONDARY OBJECTIVES:

I. To evaluate the overall response (OR) rate. II. To evaluate the progression-free survival and overall survival. III. To assess serial minimal residual disease (MRD) using clonoseq, circulating tumor deoxyribonucleic acid (ct-DNA) based serial clonal evolution.

IV. Perform baseline genomic profiling for recognizing the predictive signature for response, serial MCL specific analytes assessments while on therapy.

EXPLORATORY OBJECTIVES:

I. Clonal evolution with targeted sequencing (seq) on ctDNA samples in sequential samples using a MCL specific customized gene panel would be assessed.

II. MRD assay using IgH clonoseq and ctDNA analysis, flow cytometry at various time points from peripheral blood (PB)/bone marrow (BM).

III. Sequential immunologic studies with cytokines/chemokines using a analyte panel, T cell numbers, and immunoglobulins (Ig).

IV. Tissue microenvironmental studies with simultaneous assessment of PB, BM and lymph nodes for gene expression profiling (GEP), single cell seq, ribonucleic acid (RNA) seq and clonal heterogeneity and the impact of acalabrutinib (A)-rituximab (R) treatment.

V. Extensive bioinformatics studies. VI. Identification of signaling pathways or biomarkers that predict sensitivity after therapy.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab intravenously (IV) over 3-4 hours on days 1, 8, 15, and 22 of cycle 1, and day 1 of cycles 2-12, 14, 16, 18, 20, 22 and 24. Cycles repeats every 28 days for up to 24 months or until complete remission is achieved in the absence of disease progression or unacceptable toxicity.

After completion of study intervention, patients are followed up at 30 days for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

The study will enroll 50 elderly (≥65 years) previously untreated patient with newly diagnosed MCL.

1. Pathology confirmed diagnosis of mantle cell lymphoma with CD20 positivity and chromosome translocation t (11;14), (q13;q32) and/or positive cyclin D1 in tissue biopsy (See Appendix I, footnote 10). Cyclin D1 negative MCL are allowed after confirming the diagnosis of MCL from hem-path at MDACC.
2. Newly diagnosed elderly MCL (age ≥65 years) with no prior therapy under all risk categories
3. Patients with preexisting well-controlled cardio-vascular comorbidities - patients on anticoagulants (excluding warfarin and vitamin K antagonists), antiplatelet, anti-hypertensive, prior ablation, anti-arrhythmia, prior arrhythmias, baseline EKG abnormalities and cardiology clearance are allowed. Ejection fraction >=50% and cardiology clearance are required. (Echo and EKG and cardiology consultation within 2 months prior to C1D1 are allowed).
4. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.
5. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).
6. Bi-dimensional measurable disease using the Cheson criteria (Measurable disease by PET-CT scan defined as at least 1 lesion that measures ≥ 1.5 cm in single dimension.) Gastrointestinal, bone marrow or spleen only patients are allowable.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
8. An absolute neutrophil count (ANC) > 1,000/mm3 and platelet count >100,000/mm3 (Patients who have bone marrow and spleen infiltration by MCL are eligible, the ANC and platelets counts will not be limited).
9. Serum bilirubin <1.5 mg/dl and creatinine clearance minimum to 50 mL/min per the Cockcroft-Gault formula (Appendix VII)
10. AST (SGOT) and ALT (SGPT) < 2. x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. Gilbert's disease is allowed.
11. Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated with life expectancy of > 3 years. PI can use clinical judgement in the best interest of patients.
12. WOBP and males must be willing to use highly effective methods of birth control. therapy. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib tablet and for 12 months following the last dose of rituximab. For male subjects with a pregnant or non-pregnant WOCBP partner, should use barrier contraception, during treatment and for 2 days after the last dose of acalabrutinib and for 1 month following the last dose of rituximab even if they have had a successful vasectomy. Male subjects must agree to refrain from sperm donation during the study. (See Appendix VI)

Exclusion Criteria:

1. Prior treatment with acalabrutinib or any treatment for MCL.
2. History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

   a. Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study.

   b. Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which subject is disease-free for ≥3 years without further treatment.
3. Patients with central nervous system involvement with mantle cell lymphoma or with suspected or confirmed progressive multifocal leukoencephalopathy (PML) are excluded since those patients have very poor prognosis, need aggressive intensive chemoimmunotherapy and intrathecal chemotherapy along with BTK inhibitors and these patients would not be eligible for this study.
4. Pregnant or breast-feeding females.
5. Refractory nausea and vomiting, inability to swallow the formulated product, or malabsorption syndrome; chronic gastrointestinal disease, gastric restrictions, or bariatric surgery such as gastric bypass; partial or complete bowel obstruction, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of study treatment
6. Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components.
7. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
8. Concurrent participation in another therapeutic clinical trial.
9. Immunization with live vaccine within 4 weeks of and during therapy with Rituximab.
10. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML)
11. Any active significant infection (e.g., bacterial, viral or fungal, including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR]).
12. Serologic status reflecting active hepatitis B or C infection.

    1. Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before randomization and must be willing to undergo DNA PCR testing during the study. Those who are HbsAg-positive or hepatitis B PCR positive will be excluded.
    2. Subjects who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.13. Major surgical procedure within 30 days before the first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.

14. Patients with HIV/AIDS

15. Active bleeding, history of bleeding diathesis (such as Hemophilia or Von-Willebrand disease), Any history of intracranial bleed or stroke within 6 months of first dose of study drug.

16. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).

17. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before first dose of study drug.

18. Major surgical procedure within 30 days before the first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.

19. Requires anticoagulation with warfarin or equivalent vitamin K antagonist.

20. Concomitant use of corticosteroids at > 20 mg prednisone or equivalent per day > 2 weeks.

21. Requires treatment with strong CYP3A inhibitors or inducers (refer to section 8.6.1 and list in Appendix V).

22. Patients who have had a stroke within 6 months.

23. Any of the following conditions considered clinically significant cardiovascular diseases as determined after cardiology consultation: Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll on study.

• Diagnosed Congestive heart failure,

* Active/symptomatic coronary artery disease
* Congestive heart failure
* Myocardial infarction in the preceding 6 months,
* Significant conduction abnormalities, including but not limited to:

  o Left bundle branch block,

  o 2nd degree AV block type II,

  o 3rd degree block,

  o QT prolongation (QTc > 480 msec),

  o Sick sinus syndrome

  o Ventricular tachycardia
  * Symptomatic bradycardia (heart rate < 50 bpm),
  * Persistent, controlled and uncontrolled atrial fibrillation.
* Uncontrolled hypertension
* Hypotension,
* light headedness and syncope,

  24. Active infection

  25. Acute infection requiring systemic anti-microbial treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to initiation of therapy.

  26. Active infection including systemic fungal or CMV infection who were hospitalized in past 6 months.

  27. Any other serious medical condition including, but not limited to, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, uncontrolled hypertension i.e. Uncontrolled BP - >160/110 despite 3 different classes of full dose anti-hypertensives medications and in spite of cardiology evaluation. Documentation from cardiology is required to say that the BP is uncontrollable.), COPD, renal failure, psychiatric illness or social circumstances that, in the investigator's opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form or complying with study procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | At 16 weeks
Incidence of adverse events (AEs) | Up to 30 days following the last dose of study drug
  Toxicity is defined as all related grade 3 or higher AEs and not only the non-hematologic AEs will be considered toxicities treatment-related grade 3 or higher AEs within the first three cycles, and any treatment-related toxicities, which cause drug delays for more than 4 weeks. Toxicity data by type and severity will be summarized by frequency tables for all patients by Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Overall response rate | Up to 7 years
  Summary statistics including mean, standard deviation, median, and range for continuous variables, frequency count and percentage categorical variables will be reported. Complete response rate and its posterior credibility interval will be calculated. Response rate and its 95% confidence interval will be estimated. Logistic regression model may be fitted to assess the effects of important patient prognostic factors on response.
Progression free survival (PFS) | From the start of the treatment to progression or death due to any cause whichever happened first, assessed up to 7 years
  Estimated using Kaplan and Meier method. The log-rank test will be used to evaluate the difference in PFS between patient groups.
Overall survival (OS) | From the start of the treatment to death due to any cause, assessed up to 7 years
  Estimated using Kaplan and Meier method. The log-rank test will be used to evaluate the difference in OS between patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org